CLINICAL TRIAL: NCT02013791
Title: A Phase 2, Multi-center, Vehicle- and Sham-controlled, Randomized Study of RESTASIS® X in Patients With Moderate to Severe Dry Eye Disease
Brief Title: Phase 2 Study of a New Ophthalmic Formulation of Cyclosporine (Restasis® X) in Patients With Dry Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192371-024
Record Dates: First submitted 2013-12-12; First posted 2013-12-17 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Stage 1 Cohort 1 (Other): Vehicle administered to study eye and Sham administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Other: Sham
- Stage 1 Cohort 2 (Experimental): Cyclosporine New Ophthalmic Formulation Dose A administered to study eye and Vehicle administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 3 (Experimental): Cyclosporine New Ophthalmic Formulation Dose B administered to study eye and Vehicle administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 4 (Experimental): Cyclosporine New Ophthalmic Formulation Dose C administered to study eye and Vehicle administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 5A (Experimental): Cyclosporine New Ophthalmic Formulation Dose D administered to the study eye and vehicle administered to the non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 6A (Experimental): Cyclosporine New Ophthalmic Formulation Dose E administered to study eye and Vehicle administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 6B (Experimental): Cyclosporine New Ophthalmic Formulation Dose F administered to study eye and Vehicle administered to non-study eye on Day 1.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 6C (Experimental): Cyclosporine New Ophthalmic Formulation Dose C administered to study eye and Vehicle administered to non-study eye on Day 1 and retreatment at Week 12 if applicable.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation
- Stage 1 Cohort 6D (Experimental): Cyclosporine New Ophthalmic Formulation Dose F administered to study eye and Vehicle administered to non-study eye on Day 1 and retreatment at Week 12 if applicable.
  Interventions: Drug: Vehicle; Drug: Cyclosporine New Ophthalmic Formulation

INTERVENTIONS:
Drug: Vehicle — Vehicle of cyclosporine administered as per protocol
Other: Sham — Sham administered to non-study eye as per protocol on Day 1
  Arms: Stage 1 Cohort 1
Drug: Cyclosporine New Ophthalmic Formulation — Cyclosporine New Ophthalmic Formulation administered as per protocol
  Other Names: RESTASIS® X
  Arms: Stage 1 Cohort 2; Stage 1 Cohort 3; Stage 1 Cohort 4; Stage 1 Cohort 5A; Stage 1 Cohort 6A; Stage 1 Cohort 6B; Stage 1 Cohort 6C; Stage 1 Cohort 6D

SUMMARY:
This study will evaluate a new ophthalmic formulation of cyclosporine (Restasis® X) in patients with moderate to severe dry eye disease in two stages. Up to 3 doses will be studied in Stage 2 based on results from Stage 1. No patients participating in Stage 1 will participate in Stage 2 of this study. This study was terminated and Stage 2 of the study was cancelled.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe dry eye disease in both eyes
* Best-corrected visual acuity (BCVA) of 20/100 or better in each eye

Exclusion Criteria:

* Use of any cyclosporine preparations within 3 months
* Use of topical medications, other than artificial tears, in the eyes within 1 month
* Use of contact lenses in either eye within 1 month
* Stage 2 only: Participation in Stage 1 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Safyan, Study Director — Allergan
Locations (8):
- United States (8):
  - Sall Research Medical Center, Artesia, California
  - Lugene Eye Institute, Glendale, California
  - Lakeside Vision Center, Irvine, California
  - Steve Yoelin MD Medical Asscociates, Newport Beach, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Vision Institute, Colorado Springs, Colorado
  - Johns Hopkins University - Wilmer Eye Institute, Baltimore, Maryland
  - Eye Centers of Racine and Kenosha, Kenosha, Wisconsin

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated. Stage 2 of the study was not conducted.
Period: Period 1
Arm/Group | Stage 1 Cohort 5A | Stage 1 Cohort 4 | Stage 1 Cohort 6C | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 6B | Stage 1 Cohort 6D | Stage 1 Cohort 6A | Stage 1 Cohort 1
Started | 8 | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 3
Completed | 8 | 6 | 4 | 7 | 4 | 8 | 3 | 7 | 3
Not Completed | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Other Miscellaneous Reasons | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Stage 1 Cohort 5A | Stage 1 Cohort 4 | Stage 1 Cohort 6C | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 6B | Stage 1 Cohort 6D | Stage 1 Cohort 6A | Stage 1 Cohort 1
Started | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cohort 5A | Stage 1 Cohort 4 | Stage 1 Cohort 6C | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 6B | Stage 1 Cohort 6D | Stage 1 Cohort 6A | Stage 1 Cohort 1 | Total
Number analyzed (Participants) | 8 | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 3 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.47) | 55.3 (6.58) | 58.5 (6.95) | 50.1 (15.06) | 52.3 (11.64) | 57.4 (10.69) | 52.8 (13.45) | 53.1 (12.19) | 56.0 (7.55) | 54.0 (11.19)
Age, Customized [Count of Participants; unit: Participants]
  <45 years | 2 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 10
  45 to 65 years | 5 | 7 | 3 | 5 | 2 | 5 | 1 | 5 | 3 | 36
  >65 years | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 3 | 5 | 3 | 6 | 1 | 7 | 2 | 40
  Male | 2 | 1 | 1 | 3 | 1 | 2 | 3 | 1 | 1 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 10
  Black | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4
  Asian | 0 | 1 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 8
  Hispanic | 7 | 6 | 1 | 2 | 2 | 3 | 3 | 7 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are AEs with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to up to 24 Weeks
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 5A | Stage 1 Cohort 4 | Stage 1 Cohort 6C | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 6B | Stage 1 Cohort 6D | Stage 1 Cohort 6A | Stage 1 Cohort 1
Number analyzed (Participants) | 8 | 8 | 4 | 8 | 4 | 8 | 4 | 8 | 3
Participants | 7 | 8 | 4 | 6 | 4 | 7 | 3 | 5 | 3

2. Other Pre Specified Outcome: Change From Baseline in Corneal Staining Score Using a 6-Point Scale
Description: Total corneal staining with sodium fluorescein was measured in the study eye using the 6-point Oxford scale [Grade 0: <2 dots (best), Grade 1: ≥2 to ≤10 dots, Grade 2: >10 to ≤32 dots, Grade 3: >32 to ≤100 dots, Grade 4: >100 to ≤316 dots and Grade 5: >316 dots or ulcer/erosion (worst)]. The study eye was defined as the eye that received the dosing level of the treatment received. A negative change from Baseline represents a decrease in staining (improvement).
  Corneal Staining Score was originally registered as a Primary endpoint but it is actually an exploratory endpoint.
Time Frame: Baseline (Day 1) to Week 12
Population: Modified Intent-to-treat (mITT) Population included all participant who received study treatment and had Baseline and at least 1 post-baseline assessment. Analyses includes participants who had data at both Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 Cohort 4
Number analyzed (Participants) | 6
score on a scale
  Baseline | 2.5 (0.55)
  Change from Baseline to Week 12 | -0.8 (1.33)

ADVERSE EVENTS:
Time Frame: First dose of study drug to up to 24 Weeks
Arm/Group | Stage 1 Cohort 5A | Stage 1 Cohort 4 | Stage 1 Cohort 6C | Stage 1 Cohort 3 | Stage 1 Cohort 2 | Stage 1 Cohort 6B | Stage 1 Cohort 6D | Stage 1 Cohort 6A | Stage 1 Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/4 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8 | 4/4 | 6/8 | 4/4 | 7/8 | 3/4 | 5/8 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Cohort 5A (N=8) | Stage 1 Cohort 4 (N=8) | Stage 1 Cohort 6C (N=4) | Stage 1 Cohort 3 (N=8) | Stage 1 Cohort 2 (N=4) | Stage 1 Cohort 6B (N=8) | Stage 1 Cohort 6D (N=4) | Stage 1 Cohort 6A (N=8) | Stage 1 Cohort 1 (N=3)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Cohort 5A (N=8) | Stage 1 Cohort 4 (N=8) | Stage 1 Cohort 6C (N=4) | Stage 1 Cohort 3 (N=8) | Stage 1 Cohort 2 (N=4) | Stage 1 Cohort 6B (N=8) | Stage 1 Cohort 6D (N=4) | Stage 1 Cohort 6A (N=8) | Stage 1 Cohort 1 (N=3)
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0
Corneal deposits (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 3 | 3 | 0 | 4 | 1 | 2 | 1 | 2 | 2
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meibomian gland discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 4 | 5 | 4 | 2 | 3 | 6 | 2 | 2 | 1
Injection site pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Instillation site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Antinuclear antibody positive (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02013791/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02013791/SAP_001.pdf